CLINICAL TRIAL: NCT03573596
Title: Persistence Of Major Molecular Remission In Chronic Myeloid Leukemia After A Second Stop Of Tki Treatment In Patients Who Failed An Initial Stop Attempt: A Multicenter Prospective Trial
Brief Title: Persistence of MR3 in Chronic Myeloid Leukemia (CML) After a 2nd Stop of TKI Treatment
Acronym: DASTOP2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Uppsala University Hospital (Other); Skane University Hospital (Other); Helsinki University Central Hospital (Other); Odense University Hospital (Other); Henri Mondor University Hospital (Other); St. Olavs Hospital (Other); Helse Stavanger HF (Other Government); Aarhus University Hospital (Other); University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, J.J.W.M. Janssen, Clinical Hematologist, Deputy Chief of Department of Hematology, Amsterdam UMC, location VUmc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DASTOP2
Record Dates: First submitted 2018-05-22; First posted 2018-06-29 (Actual); Last update posted 2018-06-29 (Actual); Status verified 2018-06

CONDITIONS: CML, Relapsed
Keywords: CML; second stop; dasatinib
MeSH Terms: conditions — Recurrence | interventions — Dasatinib

STUDY DESIGN:
Intervention Model Description: Phase 2, multicenter study, prospective, open label, uncontrolled.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- dasatinib (Other): 2 years of dasatinib treatment before discontinuation if MR 4 is achieved for at least 1 year
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib — CML patients who have failed a first stopping attempt and have used any TKI for one year will switch to dasatinib 100 mg qd for an additional 2 years before second stop attempt.

SUMMARY:
This study will enroll CML patients who have failed a first TKI stopping attempt. After failure and at least a year of TKI treatment, patients will proceed to dasatinib treatment for another 2 years. If MR4 or better is re-achieved and maintained for at least one year, patients will be eligible for a second stop. After verification of MR4, TKI treatment will be stopped and patients followed in the same manner as after first stop. If MMR is lost (BCR-ABL >0.1% (IS)), TKI treatment will once again be restarted.

DETAILED DESCRIPTION:
The DASTOP2 study aims to retreat patients who relapse in the Euro-SKI study (or who stopped TKI treatment outside trials but according to EURO-SKI procedures), with TKI for at least another 3 years, out of last two years with dasatinib. If MR4 or better is re-achieved and maintained for at least one year, patients will be eligible for a second stop. After verification of MR4, TKI treatment will be stopped and patients followed in the same manner as after first stop. If MMR is lost (BCR-ABL >0.1% (IS)), TKI treatment will once again be restarted.

Patients exhibiting hematological relapse after first stop attempt will not be offered a second stop within this study. The same applies to patients in whom TKI was restarted prematurely (without loss of MMR).

ELIGIBILITY:
Inclusion Criteria:

1. CML in chronical phase (CP) under TKI treatment after failing a prior attempt to stop treatment within EURO-SKI or outside the study but according to EURO-SKI trial procedures. For the latter group this requires at least 3 years of TKI treatment (first line or second line due to intolerance to first line) before first stop, and MR4 for at least one year before stopping.
2. Treated with TKI for at least one year after having failed a prior attempt to stop TKI. Previous TKI can be any.
3. Typical BCR/ABL1 transcript (b3a2 and/or b2a2) must have been confirmed at diagnosis or later during the disease course.
4. 18 years or older.

Exclusion Criteria:

1. Previous hematological relapse after first stop of TKI.
2. Previous AP/BC at any time in the history of the disease.
3. Restart of TKI without loss of MMR after first stop
4. Current participation in another clinical study.
5. Previous or planned allogeneic stem cell transplantation.
6. Patients with contra-indications to dasatinib therapy due to comorbidities.
7. Subjects with acute hepatitis B virus (HBV) infections.
8. Uncontrolled or significant cardiovascular disease.
9. Pulmonary arterial hypertension.
10. Pleural or pericardial effusions of any grade at study entry are excluded
11. History of significant bleeding disorder unrelated to CML
12. Hypersensitivity to dasatinib and excipients of dasatinib tablets.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2018-02-01 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
successful MMR maintenance | one year
  The proportion of patients maintaining MMR at 12 months after discontinuing TKI a second time (survival without loss of major molecular response, MMR, defined as BCR-ABL1 > 0.1% on IS at one time point).

SECONDARY OUTCOMES:
correlates with succesful stop | 1 year
  Assessment of clinical and biological factors correlating with persistence of MMR or better after second TKI stop.
reachievement of MR4 | 1 year
  Number of patients who re-achieved stable MR4, and were offered study participation.
Time to reachievement of MR4 | 1 year
  Time to reachievement of MR4 after second loss of MMR.
Adverse events after TKI withdrawal | 1 year
  Adverse events related to second TKI stop, clinical and biological factors correlated to development of these AEs.
Overall survival | 1 year
  Overall survival
Progression-free survival | 1 year
  Progression-free survival
TKI restart without prior molecular relapse | 1 year
  Occurrence of a restart of TKI without prior molecular relapse.

CONTACTS AND LOCATIONS:
Overall Officials: Ulla Olsson-Strömberg, MD PhD, Principal Investigator — Department of Hematology, Uppsala University Hospital, Uppsala, Sweden
Locations (21):
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Odense University Hospital, Odense
- Helsinki University Hospital, Helsinki, Finland
- Centre Hospitalo-Universitaire, Créteil, France
- University Hospital, Bonn, Germany
- Netherlands (4):
  - VU University medical center, Amsterdam
  - Albert Schweitzer Hospital, Dordrecht
  - Radboud University medical center, Nijmegen
  - Erasmus University medical center, Rotterdam
- Norway (5):
  - Haukeland, Bergen University Hospital, Bergen
  - Oslo University Hospital, Oslo
  - Stavanger University Hospital, Stavanger
  - Tromsø University Hospital, Tromsø
  - St Olavs Hospital-Trondheim University Hospital, Trondheim
- Sweden (7):
  - University Hospital, Linköping
  - Sunderby Sjukhus, Luleå
  - Lund University Hospital, Lund
  - Örebro University Hospital, Örebro
  - Karolinska Hospital, Stockholm
  - Umeå University Hospital, Umeå
  - Uppsala University Hospital (Akademiska), Uppsala

IPD SHARING:
Plan to Share IPD: Undecided
Study results will be published as soon as possible. Steering committee will decide on sharing IPD. This is still pending.

REFERENCES:
- [Derived] Flygt H, Soderlund S, Richter J, Saussele S, Koskenvesa P, Stenke L, Mustjoki S, Dimitrijevic A, Stentoft J, Majeed W, Roy L, Wolf D, Dreimane A, Gjertsen BT, Gedde-Dahl T, Ahlstrand E, Markevarn B, Hjorth-Hansen H, Janssen J, Olsson-Stromberg U. Treatment-free remission after a second TKI discontinuation attempt in patients with Chronic Myeloid Leukemia re-treated with dasatinib - interim results from the DAstop2 trial. Leukemia. 2024 Apr;38(4):781-787. doi: 10.1038/s41375-024-02145-6. Epub 2024 Jan 26. PMID 38278960